CLINICAL TRIAL: NCT03968419
Title: A Randomized, Open-label, Phase II Study of Canakinumab or Pembrolizumab as Monotherapy or in Combination as Neoadjuvant Therapy in Subjects With Resectable Non-small Cell Lung Cancer (CANOPY-N)
Brief Title: This Study Will Evaluate the Effect of Canakinumab or Pembrolizumab Given as Monotherapy or in Combination as Neo-adjuvant Treatment for Subjects With Early Stages NSCLC.
Acronym: CANOPY-N
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study early terminated due to low enrollment compared to the anticipated figures.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885V2201C; 2018-004813-42 (EudraCT Number)
Record Dates: First submitted 2019-05-15; First posted 2019-05-30 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: ACZ885; canakinumab; pembrolizumab; NSCLC; non-small cell lung cancer; non small cell lung cancer; early stage NSCLC; squamous; non-squamous,; MPR; major pathological response; hs-CRP; PD-L1; hsCRP; surgery; neo-adjuvant; neo adjuvant; CD8; hs-IL-6; CANOPY
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — canakinumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Canakinumab monotherapy (Experimental): Participants received 200 mg of canakinumab once every 3 weeks for a maximum duration of 6 weeks prior to surgery
  Interventions: Drug: Canakinumab
- Canakinumab + pembrolizumab (Experimental): Participants received 200 mg of canakinumab in combination with 200 mg of pembrolizumab once every 3 weeks for a maximum duration of 6 weeks prior to surgery
  Interventions: Drug: Canakinumab; Drug: Pembrolizumab
- Pembrolizumab monotherapy (Experimental): Participants received 200 mg of pembrolizumab every 3 weeks for a maximum duration of 6 weeks prior to surgery
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Canakinumab — 200 mg of canakinumab administered via subcutaneous injections once every 3 weeks for a maximum duration of 6 weeks
  Other Names: ACZ885
  Arms: Canakinumab + pembrolizumab; Canakinumab monotherapy
Drug: Pembrolizumab — 200 mg of pembrolizumab administered via infusion once every 3 weeks for a maximum duration of 6 weeks
  Arms: Canakinumab + pembrolizumab; Pembrolizumab monotherapy

SUMMARY:
The purpose of this study was to evaluate the major pathological response (MPR) rate of canakinumab given as a neoadjuvant treatment, either as single agent or in combination with pembrolizumab, in addition to evaluate the MPR of pembrolizumab as a single agent and the dynamic of the tumor microenvironment changes on treatment.

DETAILED DESCRIPTION:
This was a randomized, phase II, open-label study evaluating canakinumab, an anti-IL-1β monoclonal antibody, or pembrolizumab, a monoclonal antibody designed to block the PD-1 receptor, as monotherapy or in combination as neoadjuvant therapy. The study population included adult subjects with resectable non-small cell lung cancer (NSCLC) planned for surgery in approximately 4-6 weeks. Subjects were treated for a maximum duration of 6 weeks (2 cycles) until surgery, progression, unacceptable toxicity or discontinuation from the study treatment for any other reason.

Subjects were randomized in a 2:2:1 ratio to one of the 3 treatment arms (canakinumab alone or canakinumab in combination with pembrolizumab or pembrolizumab alone). Surgery was performed between 4 to 6 weeks after the first dose of study treatment.

All randomized subjects were followed for safety for up to 130 days following the last dose of study treatment (safety follow-up period).

ELIGIBILITY:
Key inclusion criteria:

* Histologically confirmed NSCLC stage IB-IIIA (per AJCC 8th edition), deemed suitable for primary resection by treating surgeon, except for N2 and T4 tumors.
* Subject must have been eligible for surgery and with a planned surgical resection in approximately 4-6 weeks (after the first dose of study treatment).
* A mandatory newly obtained tissue biopsy from primary site was required for study enrollment. An archival biopsy was also acceptable if obtained up to 5 months before first day of study treatment and if the subject did not go through antineoplastic systemic therapies between biopsy collection date and beginning of study treatment.
* Eastern Cooperative oncology group (ECOG) performance status of 0 or 1.

Key exclusion criteria:

* Subjects with unresectable or metastatic disease.
* History of severe hypersensitivity reactions to monoclonal antibodies, which in the opinion of the investigator may pose an increased risk of serious infusion reaction
* Subjects who received prior systemic therapy (including chemotherapy, other anti-cancer therapies and any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways) in the past 3 years before screening
* Active autoimmune disease that has required systemic treatment in the past 2 years prior to randomization. Control of the disorder with replacement therapy was permitted
* Subject with suspected or proven immunocompromised state or infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- United States (4):
  - UCLA Oncology Hematology, La Jolla, California
  - University of Kansas Medical Center Neurology Dept., Kansas City, Kansas
  - SUNY - Upstate Medical University, Syracuse, New York
  - Methodist Hospital / Methodist Cancer Center, Houston, Texas
- Novartis Investigative Site, Brussels, Belgium
- Novartis Investigative Site, Montreal, Quebec, Canada
- France (3):
  - Novartis Investigative Site, Montpellier, Herault
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Paris
- Germany (4):
  - Novartis Investigative Site, Bad Berka
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, Halle
- Novartis Investigative Site, Thessaloniki, Greece
- Novartis Investigative Site, Kashiwa, Chiba, Japan
- Netherlands (3):
  - Novartis Investigative Site, 's-Hertogenbosch
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Maastricht
- Russia (2):
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Saint Petersburg
- Spain (3):
  - Novartis Investigative Site, Jaén, Andalusia
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Taipei, Taiwan
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Sakarya
  - Novartis Investigative Site, Sihhiye / Ankara

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Garrido P, Pujol JL, Kim ES, Lee JM, Tsuboi M, Gomez-Rueda A, Benito A, Moreno N, Gorospe L, Dong T, Blin C, Rodrik-Outmezguine V, Passos VQ, Mok TS. Canakinumab with and without pembrolizumab in patients with resectable non-small-cell lung cancer: CANOPY-N study design. Future Oncol. 2021 Apr;17(12):1459-1472. doi: 10.2217/fon-2020-1098. Epub 2021 Mar 2. PMID 33648347
- See also: Plain Language Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1547

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 29 centers across 12 countries.
Pre-assignment Details: Screening assessments were done within 28 days prior to randomization. A total of 163 participants were screened. Of them, 88 participants were randomized. After treatment completion or discontinuation, all subjects were followed for safety for up to 130 days following the last dose of study treatment (safety follow-up period).
Period: Treatment Period
Arm/Group | Canakinumab Monotherapy | Canakinumab + Pembrolizumab | Pembrolizumab Monotherapy
Started | 35 | 35 | 18
Completed | 35 | 35 | 17
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Period: Safety Follow-up Period
Arm/Group | Canakinumab Monotherapy | Canakinumab + Pembrolizumab | Pembrolizumab Monotherapy
Started | 35 | 35 | 18
Completed | 30 | 32 | 17
Not Completed | 5 | 3 | 1
Not completed — Death | 3 | 2 | 1
Not completed — Subject Decision | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab Monotherapy | Canakinumab + Pembrolizumab | Pembrolizumab Monotherapy | Total
Number analyzed (Participants) | 35 | 35 | 18 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.5 (9.88) | 67.1 (6.98) | 66.1 (5.61) | 66.2 (7.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 9 | 36
  Male | 22 | 21 | 9 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20 | 25 | 12 | 57
  Asian | 7 | 3 | 2 | 12
  Black or African American | 1 | 1 | 0 | 2
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Unknown | 7 | 5 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Major Pathological Response (MPR) Rate at the Time of Surgery in Subjects Randomized to Canakinumab Monotherapy and in Combination With Pembrolizumab Based on Central Review
Description: MPR was defined as the percentage of participants with major pathological response (defined as ≤10% residual viable tumor cells on surgical samples). Any participant who had >10% residual viable cancer cells, or started new antineoplastic therapy prior to surgery, or did not have the surgery performed, or had the surgery performed but with unevaluable MPR result, was considered as a non-responder.
  MPR was assessed at the time of surgery in all subjects randomized to canakinumab monotherapy and in combination with pembrolizumab based on central review.
Time Frame: At time of surgery (up to 6 weeks after first dose of study treatment)
Population: All subjects who were randomized to canakinumab monotherapy or canakinumab in combination with pembrolizumab
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab Monotherapy | Canakinumab + Pembrolizumab
Number analyzed (Participants) | 35 | 35
Percentage of participants | 2.9 [0.07 to 14.92] | 17.1 [6.56 to 33.65]

2. Secondary Outcome: Canakinumab Antidrug Antibodies (ADA) Prevalence
Description: Canakinumab ADA prevalence at baseline was calculated as the percentage of participants who had a canakinumab ADA positive result at baseline
Time Frame: Predose (0 hour) on Day 1 of Cycle 1 (Cycle=21 days)
Population: All subjects randomized to canakinumab monotherapy or canakinumab in combination with pembrolizumab who received at least one dose of canakinumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab Monotherapy | Canakinumab + Pembrolizumab
Number analyzed (Participants) | 35 | 35
Participants | 0 | 0

3. Secondary Outcome: Canakinumab ADA Incidence
Description: Canakinumab ADA incidence on treatment was calculated as the percentage of participants who were canakinumab treatment-induced ADA positive (post-baseline ADA positive with ADA-negative sample at baseline) and canakinumab treatment-boosted ADA positive (post-baseline ADA positive with titer that is at least the fold titer change greater than the ADA-positive baseline titer)
Time Frame: From baseline (Predose on Day 1 of Cycle 1) up to 130 days after last dose of study treatment (assessed up to 24.6 weeks). Cycle = 21 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab Monotherapy | Canakinumab + Pembrolizumab
Number analyzed (Participants) | 35 | 35
Participants | 1 | 0

4. Secondary Outcome: Pembrolizumab ADA Prevalence
Description: Pembrolizumab ADA prevalence at baseline was calculated as the percentage of participants who had a pembrolizumab ADA positive result at baseline
Time Frame: Predose (0 hour) on Day 1 of Cycle 1 (Cycle = 21 days)
Population: All subjects randomized to canakinumab in combination with pembrolizumab or pembrolizumab monotherapy who received at least one dose of pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab + Pembrolizumab | Pembrolizumab Monotherapy
Number analyzed (Participants) | 35 | 18
Participants | 4 | 3

5. Secondary Outcome: Pembrolizumab ADA Incidence
Description: Pembrolizumab ADA incidence on treatment was calculated as the percentage of participants who were pembrolizumab treatment-induced ADA positive (post-baseline ADA positive with ADA-negative sample at baseline) and pembrolizumab treatment-boosted ADA positive (post-baseline ADA positive with titer that is at least the fold titer change greater than the ADA-positive baseline titer)
Time Frame: From baseline (Predose on Day 1 of Cycle 1) up to 26 days after last dose of study treatment (assessed up to 10.7 weeks). Cycle = 21 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab + Pembrolizumab | Pembrolizumab Monotherapy
Number analyzed (Participants) | 35 | 18
Participants | 3 | 4

6. Secondary Outcome: Overall Response Rate (ORR) Based on Local Investigator Assessment Using RECIST v1.1
Description: ORR is defined as the percentage of subjects with confirmed best overall response of complete response (CR) or partial response (PR), as per local investigator's assessment by RECIST 1.1.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters
Time Frame: From date of randomization to date of surgery, assessed up to 6 weeks
Population: FAS including all subjects to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab Monotherapy | Canakinumab + Pembrolizumab | Pembrolizumab Monotherapy
Number analyzed (Participants) | 35 | 35 | 18
Percentage of participants | 0 [0.00 to 10.00] | 8.6 [1.80 to 23.06] | 11.1 [1.38 to 34.71]

7. Secondary Outcome: Serum Canakinumab Concentration
Description: Canakinumab serum concentrations were determined at the specified time points.
Time Frame: Predose (0 hour) on Day 1 of Cycles 1 and 2 (Cycle =21 days)
Population: All participants who received at least one dose of canakinumab with at least one evaluable pharmacokinetic (PK) sample. Number analyzed corresponds to the number of participants with an evaluable PK sample at the specified time point
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/miliLiter (ug/mL)
Arm/Group | Canakinumab Monotherapy | Canakinumab + Pembrolizumab
Number analyzed (Participants) | 35 | 35
microgram/miliLiter (ug/mL)
  Cycle 1: number analyzed (Participants) | 35 | 34
  Cycle 1 | 0 (0) | 0 (0)
  Cycle 2: number analyzed (Participants) | 35 | 34
  Cycle 2 | 10.9 (32.9) | 10.3 (41.0)

8. Secondary Outcome: Serum Pembrolizumab Concentration
Description: Pembrolizumab serum concentrations were determined at the specified time points.
Time Frame: Predose (0 hour) and 0.5 hours post dose on Day 1 of Cycle 1 and predose on Cycle 2 (Cycle =21 days)
Population: All participants who received at least one dose of pembrolizumab with at least one evaluable PK sample. Number analyzed corresponds to the number of participants with an evaluable PK sample at the specified time point
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Canakinumab + Pembrolizumab | Pembrolizumab Monotherapy
Number analyzed (Participants) | 34 | 17
ug/mL
  Cycle 1 predose: number analyzed (Participants) | 32 | 17
  Cycle 1 predose | 0 (0) | 0 (0)
  Cyle 1 0.5 hours post dose: number analyzed (Participants) | 29 | 10
  Cyle 1 0.5 hours post dose | 65.5 (23.8) | 65.5 (19.9)
  Cycle 2 predose: number analyzed (Participants) | 32 | 16
  Cycle 2 predose | 16.0 (43.4) | 35.5 (13.7)

9. Secondary Outcome: Surgical Feasibility Rate
Description: Surgical feasibility rate was defined as the percentage of subjects who underwent surgery following study treatment.
Time Frame: Up to 6 weeks after first dose
Population: FAS including all subjects to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab Monotherapy | Canakinumab + Pembrolizumab | Pembrolizumab Monotherapy
Number analyzed (Participants) | 35 | 35 | 18
Percentage of participants | 91.4 [76.94 to 98.20] | 97.1 [85.08 to 99.93] | 100 [81.47 to 100.00]

10. Secondary Outcome: Major Pathological Response (MPR) Rate at the Time of Surgery in Subjects Randomized to Pembrolizumab Monotherapy Based on Central Review
Description: MPR was defined as the percentage of participants with major pathological response (defined as ≤10% residual viable tumor cells on surgical samples). Any participant who had >10% residual viable cancer cells, or started new antineoplastic therapy prior to surgery, or did not have the surgery performed, or had the surgery performed but with unevaluable MPR result, was considered as a non-responder.
  MPR was assessed at the time of surgery in all subjects randomized to pembrolizumab monotherapy arm based on central review.
Time Frame: At time of surgery (up to 6 weeks after first dose)
Population: All subjects who were randomized to pembrolizumab monotherapy arm
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab Monotherapy
Number analyzed (Participants) | 18
Percentage of participants | 16.7 [3.58 to 41.42]

11. Secondary Outcome: Difference in Major Pathological Response (MPR) Rate Between the Canakinumab Plus Pembrolizumab Arm and the Pembrolizumab Arm Based on Central Review
Description: MPR was defined as the percentage of participants with ≤10% residual viable tumor cells on surgical samples. MPR was assessed at the time of surgery based on central review. The difference in MPR rate between the canakinumab plus pembrolizumab arm and the pembrolizumab arm based on central review along with the Chang and Zhang confidence interval was assessed.
Time Frame: At time of surgery (up to 6 weeks after first dose of study treatment)
Population: All subjects who were randomized to canakinumab in combination with pembrolizumab or pembrolizumab monotherapy arms
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab + Pembrolizumab | Pembrolizumab Monotherapy
Number analyzed (Participants) | 35 | 18
Percentage of participants | 17.1 [6.56 to 33.65] | 16.7 [3.58 to 41.42]
Statistical Analysis 1: Comparison: Canakinumab + Pembrolizumab vs Pembrolizumab Monotherapy; Difference in MPR rate; Test type: Other; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-25.56 to 21.23]

12. Secondary Outcome: Major Pathological Response (MPR) Rate at the Time of Surgery in All Subjects Based on Local Review
Description: MPR was defined as the percentage of participants with major pathological response (defined as ≤10% residual viable tumor cells on surgical samples). Any participant who had >10% residual viable cancer cells, or started new antineoplastic therapy prior to surgery, or did not have the surgery performed, or had the surgery performed but with unevaluable MPR result, was considered as a non-responder.
  MPR was assessed at the time of surgery in all subjects based on local review.
Time Frame: At time of surgery (up to 6 weeks after first dose)
Population: FAS including all subjects to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab Monotherapy | Canakinumab + Pembrolizumab | Pembrolizumab Monotherapy
Number analyzed (Participants) | 35 | 35 | 18
Percentage of participants | 0 [0.00 to 10.00] | 20.0 [8.44 to 36.94] | 22.2 [6.41 to 47.64]

13. Secondary Outcome: Major Pathological Response (MPR) Rate Based on the Levels of Biomarkers
Description: MPR was defined as the percentage of participants with major pathological response (defined as ≤10% residual viable tumor cells on surgical samples). Any participant who had >10% residual viable cancer cells, or started new antineoplastic therapy prior to surgery, or did not have the surgery performed, or had the surgery performed but with unevaluable MPR result, was considered as a non-responder.
  MPR rate was analyzed by the biomarker subgroups at baseline. Biomarkers included PD-L1, CD8, hs-CRP and hs-IL-6.
Time Frame: From date of randomization up to 6 weeks after first dose
Population: All subjects to whom study treatment was assigned by randomization. Number analyzed is the number of participants with data available for analysis for each category
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab Monotherapy | Canakinumab + Pembrolizumab | Pembrolizumab Monotherapy
Number analyzed (Participants) | 35 | 35 | 18
Percentage of participants
  PD-L1: <1%: number analyzed (Participants) | 12 | 14 | 7
  PD-L1: <1% | 0 [0.00 to 26.46] | 7.1 [0.18 to 33.87] | 14.3 [0.36 to 57.87]
  PD-L1: 1-49%: number analyzed (Participants) | 15 | 13 | 6
  PD-L1: 1-49% | 6.7 [0.17 to 31.95] | 15.4 [1.92 to 45.45] | 16.7 [0.42 to 64.12]
  PD-L1: >=50%: number analyzed (Participants) | 6 | 7 | 3
  PD-L1: >=50% | 0 [0.00 to 45.93] | 42.9 [9.90 to 81.59] | 0 [0.00 to 70.76]
  hs-CRP: <2mg/L: number analyzed (Participants) | 8 | 13 | 8
  hs-CRP: <2mg/L | 12.5 [0.32 to 52.65] | 7.7 [0.19 to 36.03] | 37.5 [8.52 to 75.51]
  hs-CRP: >=2mg/L: number analyzed (Participants) | 26 | 22 | 9
  hs-CRP: >=2mg/L | 0 [0.0 to 13.23] | 22.7 [7.82 to 45.37] | 0 [0.00 to 33.63]
  hs-IL-6: <Q1 (2.52 mg/L): number analyzed (Participants) | 6 | 8 | 7
  hs-IL-6: <Q1 (2.52 mg/L) | 16.7 [0.42 to 64.12] | 12.5 [0.32 to 52.65] | 14.3 [0.36 to 57.87]
  hs-IL-6: >=Q1 (2.52 pg/mL) to <Q2 (5.36 pg/mL): number analyzed (Participants) | 8 | 10 | 3
  hs-IL-6: >=Q1 (2.52 pg/mL) to <Q2 (5.36 pg/mL) | 0 [0.00 to 36.94] | 10 [0.25 to 44.50] | 33.3 [0.84 to 90.57]
  hs-IL-6: >=Q2 (5.36 pg/mL) to <Q3 (12.03 pg/mL): number analyzed (Participants) | 8 | 7 | 6
  hs-IL-6: >=Q2 (5.36 pg/mL) to <Q3 (12.03 pg/mL) | 0 [0.00 to 36.94] | 28.6 [3.67 to 70.96] | 16.7 [0.42 to 64.12]
  hs-IL-6: >=Q3 (12.03 pg/mL): number analyzed (Participants) | 10 | 10 | 1
  hs-IL-6: >=Q3 (12.03 pg/mL) | 0 [0.00 to 30.85] | 20.0 [2.52 to 55.61] | 0 [0.00 to 97.50]
  CD8: <3%: number analyzed (Participants) | 12 | 23 | 5
  CD8: <3% | 0 [0.00 to 26.46] | 13.0 [2.78 to 33.59] | 0 [0.00 to 52.18]
  CD8: >=3%: number analyzed (Participants) | 18 | 9 | 6
  CD8: >=3% | 0 [0.00 to 18.53] | 22.2 [2.81 to 60.01] | 33.3 [4.33 to 77.72]

ADVERSE EVENTS:
Time Frame: From day of first dose of study medication to 130 days after last dose of study medication, up to 25.6 weeks
Description: Any sign or symptom that occurs during the study treatment plus the 130 days post treatment
Arm/Group | Canakinumab Monotherapy | Canakinumab + Pembrolizumab | Pembrolizumab Monotherapy
All-Cause Mortality (participants affected / at risk) | 3/35 | 2/35 | 1/18
Serious Adverse Events (participants affected / at risk) | 10/35 | 9/35 | 4/18
Other Adverse Events (participants affected / at risk) | 28/35 | 27/35 | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab Monotherapy (N=35) | Canakinumab + Pembrolizumab (N=35) | Pembrolizumab Monotherapy (N=18)
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 2 | 1 | 1
Endocarditis (Infections and infestations) | 1 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0
Pyopneumothorax (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab Monotherapy (N=35) | Canakinumab + Pembrolizumab (N=35) | Pembrolizumab Monotherapy (N=18)
Anaemia (Blood and lymphatic system disorders) | 9 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 5 | 1
Hypothyroidism (Endocrine disorders) | 0 | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 6 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 4 | 3 | 3
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1
Asthenia (General disorders) | 2 | 2 | 1
Chest pain (General disorders) | 2 | 2 | 1
Fatigue (General disorders) | 9 | 5 | 4
Influenza like illness (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1
Pain (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 6 | 2
Wound complication (Injury, poisoning and procedural complications) | 0 | 2 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 3 | 2
Amylase increased (Investigations) | 2 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 0
Bilirubin conjugated increased (Investigations) | 4 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 4 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 2 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 2 | 1
Lipase increased (Investigations) | 2 | 1 | 1
Lymphocyte count decreased (Investigations) | 4 | 0 | 1
SARS-CoV-2 test negative (Investigations) | 2 | 3 | 3
SARS-CoV-2 test positive (Investigations) | 2 | 1 | 1
Weight decreased (Investigations) | 1 | 1 | 1
White blood cell count decreased (Investigations) | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 4 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 2 | 1
Headache (Nervous system disorders) | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT03968419/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT03968419/SAP_001.pdf